CLINICAL TRIAL: NCT05188885
Title: A Real World, Multi-centric, Observational Registry Study of Chronic Kidney Diseases
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, XueQing Yu, Clinical Professor, Guangdong Provincial People's Hospital
Other Study IDs: GDPH-CKD-MIP-01
Record Dates: First submitted 2021-12-22; First posted 2022-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, white cells, urine, urine sediment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic kidney disease (CKD) refers to a variety of different diseases characterized by impairment of kidney structure and/or renal function. The prevalence of CKD in China is as high as 10.8%. With a population of more than 150 million, China has the largest number of CKD patients all over the world. People with CKD would not only progress to uremia and need renal replace treatment, it also significantly increases risk of cardiovascular disease than non-CKD population. It has created a heavy burden on people's health and national economy. There is an urgent need to establish an effective system for CKD prevention and control in China. Evidences from large sample cohort and real world based research are still rare. This study will provide good experience for reducing the occurrence and development of CKD.

DETAILED DESCRIPTION:
This study is designed as an investigator-initiated, multi-center, prospective and observational real world study based on mainland Chinese population. The investigators aimed to investigate the occurrence, development, treatment, prognosis state and related risk factors of CKD in China.

This study based on the standardized data network, which provides efficient data collection, integration and analysis for researchers and clinicians in multi-centers.

The sample size of this study was estimated by statisticians, epidemiologists and clinicians. Real-world studies adopted an open standard for inclusion and exclusion, larger sample size could cover a wider group of patients and take the possibility of loss of follow-up into account. Subgroup analysis can be performed in a heterogeneous population and expand the significance of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CKD as defined in the KDIGO Clinical Practice Guidelines for the Evaluation and Management of Chronic Kidney Disease 2012 Edition;
* Non-CKD patients with hypertension, diabetes, hyperlipidemia, hyperuricemia, eGFR (CKD-EPI formula) of 60-89 ml/min/1.73m^2 and other risk factors for CKD;
* Healthy population.
* Signed the informed consent voluntarily.

Exclusion Criteria:

。Patients identified to be unsuitable for enrollment by the study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrolled based on both hospitals and communities.
Sampling Method: Non-Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2021-12-27 (Actual); Primary Completion 2026-12-27 (Estimated); Study Completion 2028-12-27 (Estimated)

PRIMARY OUTCOMES:
The occurrence of chronic kidney diseases in non-CKD participants | up to 5 years
  The occurrence of chronic kidney disease is defined by KDIGO (Kidney Disease: Improving Global Outcomes) in 2012.
The progression of chronic kidney diseases in CKD participants | up to 5 years
  The progression of chronic kidney disease is defined as: Patients with baseline estimated glomerular filtration rate (eGFR) ≥60 ml /min/1.73m2 had an eGFR decrease of 30% or more, and decreased to <60 ml /min/1.73m2; Or a 50% or greater decrease in baseline eGFR <60 ml /min/1.73m2; Or end-stage renal disease (eGFR <15 ml /min/1.73m2, or initiation of renal replacement therapy)

SECONDARY OUTCOMES:
Progression in albuminuria | up to 5 years
  Progression in albuminuria: Patients with baseline urinary albumin to creatinine Ratio (uACR) <30 mg/g had uACR doubled and increased to ≥30 mg/g; or patients with baseline uACR <300 mg/g had a doubling of uACR and an increase to ≥300 mg/g.
New onset of albuminuria | up to 5 years
  Onset of albuminuria: Patients with baseline uACR <30 mg/g increased to ≥30 mg/g.
New onset of macroalbuminuria | up to 5 years
  Onset of macroalbuminuria: Patients with baseline uACR <300 mg/g increased to ≥300 mg/g.
Composite endpoints of progression of chronic kidney disease and progression of albuminuria | up to 5 years
  Composite endpoints of progression of chronic kidney disease and progression of albuminuria.
Composite endpoint of progression of chronic kidney disease, progression of albuminuria, and all-cause death. | up to 5 years
  Composite endpoint of progression of chronic kidney disease, progression of albuminuria, and all-cause death.
Change of estimated eGFR | up to 5 years
  Change rate per year.
change of uACR | up to 5 years
  Change rate per year.
Rapid decrease of renal function | up to 5 years
  The annual decrease rate of eGFR was > 5mL/min/1.73m2.

OTHER OUTCOMES:
The occurrence and development of complications of chronic renal disease | up to 5 years
  Renal anemia, renal hypertension, mineral bone metabolism disorders, etc.
Rate of Participants with cardiovascular events. | up to 5 years
  Rate of Participants with cardiovascular events.
Rate of Participants with cerebrovascular events. | up to 5 years
  Rate of Participants with cerebrovascular events.
All causes mortality | up to 5 years
  All causes mortality.
Rate of Participants with hospitalization. | up to 5 years
  Rate of Participants with hospitalization.
Changes in cognitive function score. | up to 5 years
  Changes in cognitive function score by questionnaire.
Rate of Participants with new-onset diabetes | up to 5 years
  Rate of Participants with new-onset diabetes.
Rate of Participants with severe infection | up to 5 years
  Rate of Participants with infections that need intravenous injections or hospitalization.
Rate of Participants with bone fracture | up to 5 years
  Rate of Participants with bone fracture.
Rate of Participants with tumor | up to 5 years
  Rate of Participants with tumors.
Rate of Participants with malnutrition | up to 5 years
  A decrease of body weight more than 15%, and/or serum albumin decreased to less than 30 g/L.
Rate of Participants with pregnancy | up to 5 years
  Rate of Participants with pregnancy and birth

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD, Study Chair — Guangdong Provincial People's Hospital; Zhiming Ye, MD, Study Director — Guangdong Provincial People's Hospital; Feng Wen, MD, Principal Investigator — Guangdong Provincial People's Hospital; Ting Lin, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (8):
- China (8):
  - The Second People's Hospital of Nanhai District in Foshan City, Foshan, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Wuhua County People's Hospital, Meizhou, Guangdong
  - Fogang County People's Hospital, Qingyuan, Guangdong
  - People's Hospital of Yingde, Qingyuan, Guangdong
  - Zhuhai Golden Bay Central Hospital, Zhuhai, Guangdong
  - Ganzhou Municipal Hospital, Ganzhou, Jiangxi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data that supports the results will be shared following publication. Any sub-study analysis and publication will have to be reviewed and approved by the Trial Steering Committee, local Ethics and Regulatory requirements.